CLINICAL TRIAL: NCT05118347
Title: Effects of Buteyko Breathing Technique Versus Incentive Spirometer on Breath Holding Time, Cardiopulmonary Endurance and Quality of Life in Patients With Post Lung Tumor Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahbaz Ahmad (Other)
Collaborators: University of Lahore (Other)
Responsible Party: Sponsor-Investigator, Shahbaz Ahmad, Shahbaz Ahmad, University of Lahore
Organization: University of Lahore (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SAhmadMSK
Record Dates: First submitted 2021-10-20; First posted 2021-11-12 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Lung Tumor Resuction
Keywords: Buteyko Breathing Technique; Incentive Spirometer; Control Pause; Breath Holding Time; Lung Tumor Resection

STUDY DESIGN:
Intervention Model Description: Study participants will be randomized into two groups, Buteyko breathing technique group and incentive spirometry group
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Buteyko Breathing Technique (Experimental): Buteyko Breathing Method teaches you how to bring your breathing volume back toward normal or, in other words, reverse what's called chronic hyperventilation or chronic over-breathing. When your breathing is normal (ideally it is shown you should breathe lightly, in a calm fashion, and only through the nose, not mouth), you have better oxygenation of tissues and organs, including your brain.
  Interventions: Other: Buteyko Breathing Technique
- Incentive Spirometer (Experimental): An incentive spirometer is a device that measures how deeply you can inhale (breathe in). It helps you take slow, deep breaths to expand and fill your lungs with air. This helps prevent lung problems, such as pneumonia. The incentive spirometer is made up of a breathing tube, an air chamber, and an indicator.
  Interventions: Other: Buteyko Breathing Technique

INTERVENTIONS:
Other: Buteyko Breathing Technique — An incentive spirometer is a device that measures how deeply you can inhale (breathe in). It helps you take slow, deep breaths to expand and fill your lungs with air. This helps prevent lung problems, such as pneumonia. The incentive spirometer is made up of a breathing tube, an air chamber, and an indicator.
  Other Names: Incentive Spirometer

SUMMARY:
The pulmonary complications are the major cause of morbidity and mortality following Lung surgeries. The Buteyko breathing technique is used for reversing the health condition such as poor breathing, mouth breathing and over breathing. Incentive spirometry is widely used postoperatively in the belief that intermittent ventilation restores alveolar aeration and improves oxygenation. Objective of this study will be to compare the effects of Buteyko breathing technique versus Incentive Spirometer on breath holding time, cardiopulmonary endurance and quality of life in patients with post lung tumor resection. Sample size was calculated using Control Pause as outcome measure was 16 in each group after adding 20% dropout the sample size will be 16+3=19 in each group. Participants will be randomized in to two groups Buteyko breathing technique group and incentive spirometry group. Data will be collected by the Purposive Sampling technique. Breath Holding time, cardiopulmonary endurance and quality of life will be measured for both groups at the beginning of study (1st post-operative day) and after the end of training (5th post-operative day). Data will be entered into SPSS for Statistical Analysis.

DETAILED DESCRIPTION:
The pulmonary complications are the major cause of morbidity and mortality following Lung surgeries. The Buteyko breathing technique is used for reversing the health condition such as poor breathing, mouth breathing and over breathing. Incentive spirometry is widely used postoperatively in the belief that intermittent ventilation restores alveolar aeration and improves oxygenation. Objective of this study will be to compare the effects of Buteyko breathing technique versus Incentive Spirometer on breath holding time, cardiopulmonary endurance and quality of life in patients with post lung tumor resection. Sample size was calculated using Control Pause as outcome measure was 16 in each group after adding 20% dropout the sample size will be 16+3=19 in each group. Participants will be randomized in to two groups Buteyko breathing technique group and incentive spirometry group. Data will be collected by the Purposive Sampling technique. Breath Holding time, cardiopulmonary endurance and quality of life will be measured for both groups at the beginning of study (1st post-operative day) and after the end of training (5th post-operative day). Data will be entered into SPSS for Statistical Analysis. Study will be completed within 9 months after the approval of synopsis. Participants included the study will be those who underwent lung surgery for the first time. Both male and female will be included. The patient of age between 45-55 years. Hyperventilated patient due to post-operative pain. Participants excluded were those having Post-operative renal failure or arrhythmia needed for a pacemaker. Post-operative mechanical ventilation (more than 24 hours). Patients suffering from Cardiac diseases. (Congenital heart disease, Coronary artery disease (narrowing of the arteries), Deep vein thrombosis and pulmonary embolism, Heart attack, Heart failure. And Heart muscle disease)

ELIGIBILITY:
Inclusion Criteria:

* The patients who underwent lung surgery for the first time.
* Both male and female will be included.
* The patient of age between 45-55 years.
* Hyperventilated patient due to post-operative pain

Exclusion Criteria:

* Post-operative renal failure or arrhythmia needed for a pacemaker.
* Post-operative mechanical ventilation (more than 24 hours).
* Patients suffering from Cardiac diseases. (Congenital heart disease, Coronary artery disease (narrowing of the arteries), Deep vein thrombosis and pulmonary embolism, Heart attack, Heart failure. And Heart muscle disease).

Ages: 45 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-03-15 (Estimated); Study Completion 2022-03-15 (Estimated)

PRIMARY OUTCOMES:
Breath Holding Time | 7 days
  A test used as a rough index of cardiopulmonary reserve, measured by the length of time a person can hold his or her breath after normal relaxed breathing until the slight feeling of next breath. Control Pause correlate well with the severity of disease and will be measured in seconds. Control pause is reliable and valid variable to find out the severity of disease i-e a person who can hold his breath up to 40s. It will indicate a good pulmonary condition and a person who cannot hold breath up to 10s is in status of poor pulmonary condition.
Cardiopulmonary Endurance | 7 days
  Cardiorespiratory endurance is the level at which your heart, lungs, and muscles work together when you're exercising for an extended period of time. it will be measured by 6 minutes walk test. Higher the cardiopulmonary endurance indicate a good pulmonary condition.
Quality of Life | 7 days
  World Health Organization defines Quality of Life as an individual's perception of their position in life in the context of the culture and value systems in which they live and in relation to their goals, expectations, standards and concerns. it will be measured by WHO Quality of Life Questionnaire at the scale of 0-100. 0 indicates worst quality of life and 100 indicates good quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Faiza Sharif, Principal Investigator — University of Lahore; Bilal Umer, Principal Investigator — University of Lahore
Locations (1):
- Shahbaz Ahmad, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No